CLINICAL TRIAL: NCT03535207
Title: Phase II Study of High-dose （86 Gy）Intensity Modulated Radiotherapy and Concurrent Paclitaxel and Cisplatin in Locoregionally Advanced Esophageal Cancer
Brief Title: High-dose Intensity Modulated Radiotherapy and Concurrent Chemotherapy in Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, director, department of radiation, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH201802
Record Dates: First submitted 2018-05-01; First posted 2018-05-24 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high dose chemoradiotherapy (Experimental): all eligible patients receive intensity-modulated radiotherapy 50 Gy in 25 fractions over 5 weeks and concurrent paclitaxel and cisplatin once weekly for 5 weeks，followed by hyperfractionated intensity-modulated radiotherapy boost to gross tumor volume concurrent with the same chemotherapy
  Interventions: Radiation: high dose chemoradiotherapy

INTERVENTIONS:
Radiation: high dose chemoradiotherapy — Radiation therapy: 50 Gy at 2 Gy/Fx/d on weeks 1-5,followed by 36 Gy in 30 fractions of 1.2 Gy, twice per day,on weeks 6-8 to a total dose of 86 Gy.
  concurrent chemotherapy: weekly carboplatin area under the curve (AUC) 1.5-2 and paclitaxel 45-50 mg/m2 over the duration (8 weeks) of radiation therapy.
  Adjuvant chemotherapy after high dose chemoradiation is optional.

SUMMARY:
To assess the efficacy and feasibility of high-dose intensity-modulated radiotherapy with concurrent weekly paclitaxel and cisplatin for patients with locoregionally advanced esophageal cancer

DETAILED DESCRIPTION:
The Radiation Therapy Oncology Group (RTOG) 8501 has established concurrent radiochemotherapy as the standard of care for cancer of the esophagus.However, locoregional failure remains problematic, with 25% of patients having persistence and 20% relapse of locoregional disease following the standard dose (50-50.4 Gy) chemoradiotherapy . Our previous phase I radiation dose escalation trial established the maximum tolerated dose of 86 Gy with concurrent weekly paclitaxel and cisplatin in advanced esophageal cancer.The aim of this phase II study is to examine the efficacy of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary squamous cell carcinoma of the esophagus
* Age 1 8-75.
* Patients must be deemed unresectable disease or patient is not deemed operable due to medical reasons.
* Eastern Cooperative Oncology Group （ECOG） performance status 0 to 2
* No prior radiation to the thorax that would overlap with the current treatment field.
* Patients with nodal involvement are eligible
* Adequate bone marrow, renal and hepatic functions as assessed by the following: Hemoglobin >/= 10.0 g/dl, Platelet count >/= 1 00,000/ mm^3,absolute granulocyte count (AGC) ≥2 × 10^9 cells/L,bilirubin and Aspartate transaminase ≤1.5 ×upper limit of normal (ULN), Creatinine </ =1 .5 times ULN.
* A signed informed consent must be obtained prior to therapy.
* Induction chemotherapy is allowed

Exclusion Criteria:

* The presence of a fistula.
* Prior radiotherapy that would overlap the radiation fields.
* gastroesophageal junction cancer or the lower third esophageal cancer invading the gastric wall.
* Uncontrolled concurrent illness including, but not limited to: Chronic Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness, serious uncontrolled infection, symptomatic congestive heart failure (CHF),unstable angina pectoris, uncontrolled hypertension,or psychiatric illness/social situations that would limit compliance with the study requirements.
* Known hypersensitivity to paclitaxel.
* Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
* Acquired Immune Deficiency Syndrome.
* Conditions precluding medical follow-up and protocol compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | one year
  survival time was measured from the date of study enrollment to the date of death or last follow-up

SECONDARY OUTCOMES:
toxicities | 1 year
  Acute toxicities were graded according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTC) version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Tingfeng Chen, MD, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Genernal Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herskovic A, Martz K, al-Sarraf M, Leichman L, Brindle J, Vaitkevicius V, Cooper J, Byhardt R, Davis L, Emami B. Combined chemotherapy and radiotherapy compared with radiotherapy alone in patients with cancer of the esophagus. N Engl J Med. 1992 Jun 11;326(24):1593-8. doi: 10.1056/NEJM199206113262403. PMID 1584260
- [Result] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156